CLINICAL TRIAL: NCT05067725
Title: Evaluating the Effectiveness of Migraine CarePath
Brief Title: Evaluating the Effectiveness of a Headache Management Program in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Apoorva Pradhan, Staff Scientist, Geisinger Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-0729
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Headache, Migraine; Headache
Keywords: Clinical care evaluation; Primary care
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Prospective cluster randomized control study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of practice
- CarePath Intervention (Experimental): Clinician decision support computer tool that consists of a best practice alert (BPA) embedded with a headache questionnaire, Medication Express Lane (for medication ordering), and Ask-a-doc button (for prompt virtual consultation with a neurologist)
  Interventions: Other: CarePath

INTERVENTIONS:
Other: CarePath — During an in-clinic patient encounter with a primary care provider (PCP) in any one of the intervention CMSL sites, the BPA is fired when any type of headache or migraine is entered as a diagnosis or chief complaint. The purpose of the headache assessment questionnaire is to assist the PCP in characterizing patients' headache. The Express Lane will help guide PCP decision-making for prescribing medications, lab/image ordering, and referrals. The Ask-a-doc button will provide timely access to a virtual treatment and diagnosis consult with a neurologist.
  Arms: CarePath Intervention

SUMMARY:
Between January 2020 to August 2021, fifty percent of patients referred from Geisinger's primary care sites to Neurology for headaches did not trial appropriate first line therapy prior to referral, and there was limited access available at Geisinger's Neurology department. This project was initiated to improve patient experience, management of headache, and provider experience as it relates to headache management. Geisinger's Neurology department, pharmacy department, and Community Medicine Service Line (CMSL) sites have collaborated to develop a Headache CarePath (i.e., a best practice alert containing: an EPIC headache assessment, Express Lane for prescriptions, and Ask-a-doc button for Neurology consult) and piloted at 2 CMSL sites (Woodbine, Selinsgrove) to gain some initial feedback. The feedback has been incorporated into best practice alert (BPA) language and criteria. The project team now plans to implement this CarePath to half of CMSL sites first while the other half of CMSL sites will continue to practice the standard of care as of today. The team will evaluate the impact of this CarePath on patient outcomes [change in Headache Impact Test-6 (HIT-6) scores, change in the frequency of headaches, and change in pain intensity], emergency department (ED) visits, number of referrals to Neurology for headache, and prescribing of headache medications by comparing the measures in clinics that had the CarePath implemented to those that did not. Patient outcomes will be collected by Geisinger's Survey Core, which will reach out telephonically to patients to ask about the status of their headaches (HIT-6, frequency, intensity of headaches, M-TOQ-5). Other measures will be collected and analyzed using secondary data sources such as electronic health record (EHR) data. The initial implementation is planned for 6-9 months. The findings from this evaluation will help the CarePath team identify any remaining opportunities or guide the direction of its future enhancements of the CarePath tools. The results of this evaluation will be shared with the Geisinger leadership to demonstrate its value to the organization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age for whom the Headache BPA fires at the time for their PCP encounter
* New or returning patients with headache as visit diagnosis or chief complaint for the office visit or telemedicine encounter
* Have a minimum baseline HIT-6 score of ≥ 50 points OR
* Headache frequency of ≥ 12 days with headache or migraine complaint in the last 3 months

Exclusion Criteria:

* Patients at the pilot sites (i.e., woodbine, selinsgrove)
* Patients diagnosed with secondary headache disorders (eg, brain tumors) or serious systemic illness (eg, uncontrolled hypertension, hepatic or renal failure, cardiac failure) or acute infectious illness (eg, flu, sinusitis).
* Patients with headaches as a symptom due to fall/injury
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Headache Impact Test-6 (HIT-6) score from baseline to follow up | baseline, 3 months and 6 months post baseline
  A global measure of adverse headache impact. The final HIT-6 score is obtained from simple summation of the six items and ranges between 36 and 78, with larger scores reflecting greater impact.

SECONDARY OUTCOMES:
Change in headache frequency from baseline to follow up | baseline, 3 months and 6 months post baseline
  Headache frequency will be measured as the number of days in the last 3 months the patient experiences a headache.
Change in pain intensity score from baseline to follow up | baseline, 3 months and 6 months post baseline
  Headache pain intensity will be assessed using a visual analog scale 0 - 10, where 0=no pain at all, and 10=pain as bad as it can be.
Change in the proportion of patients who received a prescription for headache medication from baseline to follow up | baseline, 3 months and 6 months post baseline
  Proportion of patients who receive a prescription for either of the medications listed below:
  * Abortive
  * Preventative
  * CGRPi
Change in the number of emergency department visits from baseline to follow up | baseline, 3 months and 6 months post baseline
  Number of patients who experience an emergency department encounter for any of the causes listed below:
  * All-cause
  * Headache-associated
Change in the proportion of patients who received a referral to neurology for headache from baseline to follow up | baseline, 3 months and 6 months post baseline
  Proportion of patients who were referred to neurology for headache

CONTACTS AND LOCATIONS:
Overall Officials: Apoorva Pradhan, BAMS, MPH, Principal Investigator — Geisinger Clinic; Eric Wright, PharmD, MPH, Study Director — Geisinger Clinic
Locations (1):
- Geisinger Clinic, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Other researchers can request access to data collected from study participants by reaching out to the P.I.

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT05067725/SAP_000.pdf